CLINICAL TRIAL: NCT06319534
Title: A Randomized Controlled Study to Explore the Effect of Stellate Ganglion Block in Dysphagic Patients With Bulbar Palsy After Ischemic Stroke
Brief Title: Stellate Ganglion Block in Bulbar Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copka Sonpashan (Other Government)
Responsible Party: Sponsor-Investigator, Copka Sonpashan, Research Director, Chao Phya Abhaibhubejhr Hospital
Organization: Chao Phya Abhaibhubejhr Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGB-ZHENQIU
Record Dates: First submitted 2024-03-10; First posted 2024-03-20 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Bulbar Palsy
MeSH Terms: conditions — Bulbar Palsy, Progressive | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive rehabilitation+Stellate ganglion block (Experimental): Patients enrolled are firstly numbered for privacy with software and divided into the observation group and the control group with. Additionally, the staffs involved in assessment would not participate in the intervention of the study. The treatment lasts 10 days.
  Interventions: Behavioral: Comprehensive rehabilitation; Procedure: Stellate ganglion block; Drug: Lidocaine Hydrochloride
- Comprehensive rehabilitation+placebo (Placebo Comparator): Patients enrolled are firstly numbered for privacy with software and divided into the observation group and the control group with. Additionally, the staffs involved in assessment would not participate in the intervention of the study. The treatment lasts 10 days.
  Interventions: Behavioral: Comprehensive rehabilitation; Behavioral: placebo injection

INTERVENTIONS:
Behavioral: Comprehensive rehabilitation — All the participants are provided with the comprehensive rehabilitation (routine rehabilitation and swallowing function training). The routine rehabilitation included intervention for risk factors (blood pressure, blood lipids, blood glucose, smoking and alcohol restriction, exercise, etc.).
Procedure: Stellate ganglion block — The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck. The ultrasonic instrument is used to determine the position.
  Arms: Comprehensive rehabilitation+Stellate ganglion block
Drug: Lidocaine Hydrochloride — the patients are provided with Stellate ganglion block, using 2.8ml of 0.8% Lidocaine hydrochloride and 0.2 ml of 0.5% vitamin B12. The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck. The ultrasonic instrument is used to determine the position.
  Arms: Comprehensive rehabilitation+Stellate ganglion block
Behavioral: placebo injection — 2.8 milliliter of normal saline will be used for injection. The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck. The ultrasonic instrument is used to determine the position.
  Arms: Comprehensive rehabilitation+placebo

SUMMARY:
This is a randomized controlled study, including dysphagic patients with bulbar palsy after ischemic stroke who were received in the department of rehabilitation medicine in 3 hospitals in China. All patients are randomly allocated to the observation group or the control group. Both groups are provided with comprehensive rehabilitation. Besides, the observation group additionally undergoes the stellate ganglion block. At admission and after 10-day treatment, video fluoroscopic swallowing study, ultrasound diagnostic devices, and penetration-aspiration scale, Flexible laryngoscope are used to assess swallowing function.

DETAILED DESCRIPTION:
Palliation of dysphagia in patients with bulbar palsy after ischemic stroke continues to be a challenge.This is a randomized controlled study, including dysphagic patients with bulbar palsy after ischemic stroke who were received in the department of rehabilitation medicine in 3 hospitals in China. All patients are randomly allocated to the observation group or the control group. Both groups are provided with comprehensive rehabilitation. Besides, the observation group additionally undergoes the stellate ganglion block. At admission and after 10-day treatment, video fluoroscopic swallowing study, and penetration-aspiration scale, ultrasound diagnostic devices, Flexible laryngoscope are used to assess swallowing function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ischemic stroke according to the diagnostic criteria, with the stroke occurring in the medulla oblongata and diagnosed as bulbar palsy.
* Age >18 years.
* First-time stroke.
* Steady vital signs,
* Transferred or admitted to the Department of Rehabilitation Medicine within 15-30d after onset.
* No cognitive impairment or aphasia, with the Montreal Cognitive Assessment score ≥21 points.
* No history of severe mental illness or psychotropic drug dependence.
* Unsafe or insufficient oral intake, indicating the need for enteral feeding

Exclusion Criteria:

* Contraindications for Stellate Ganglion Block..
* Structural abnormalities of the oropharynx.
* Complicated with other neurological diseases.
* Tracheostomy tube inserted.
* Simultaneously suffering from liver, kidney failure, tumors, or hematological diseases.
* Dysphagia caused by other possible diseases.
* Pregnant females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2024-03-23 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-07-05 (Actual)

PRIMARY OUTCOMES:
Modified Barium Swallow Impairment Profile | day 1 before any intervention, day 11, and day 60
  The Modified Barium Swallow Impairment Profile is used to evaluate the clinical severity of dysphagia. It consisted of 17 items. The total scores could range between 0 and 55, with higher scores indicating worse function.

SECONDARY OUTCOMES:
Murray secretion severity scale | day 1 before any intervention, day 11, and day 60
  Murray secretion severity scale is used for assessment of Pharyngeal secretion. The result was divided into 0-3 levels (0, normal; 1, a small amount of secretion remained and not entering the laryngeal vestibule; 2: temporary accumulation in the laryngeal vestibule; 3: persistent accumulation in the laryngeal vestibule. A higher score indicates the worse dysphagia.
Yale pharyngeal residue severity rating scale | day 1 before any intervention, day 11, and day 60
  The Yale pharyngeal residue severity rating scale was recruited for assessment of Pharyngeal residue.The result would be divided into 5 levels (1, no residue; 2, the covered pharyngeal mucosa; 3, mild residue, less than 50%; 4, moderate residue, more than 50%; 5, severe residue, spillage from laryngeal vestibule observed). A higher score indicates the worse dysphagia.
Penetration-Aspiration Scale | day 1 before any intervention, day 11, and day 60
  Penetration-Aspiration Scale was used to assess dysphagia under Videofluoroscopic Swallowing Study, primarily evaluating the extent to which fluid food entered the airway and caused penetration or aspiration during the swallowing process. As the level increased, the severity of dysphagia also increased.
Generalized Anxiety Disorder 7-item scale | day 1 before any intervention, day 11, and day 60
  Generalized Anxiety Disorder 7-item scale was used to assess anxiety.The total score could range from 0 to 21, with higher scores indicating more severe anxiety.
Movement distances of the hyoid bone | day 1 before any intervention, day 11, and day 60
  The lateral swallowing fluorography record was decomposed into individual images. Images were selected at both the resting positions and the maximum displacement. The distance of position change for the hyoid bone between the two images was measured with the inferior border of the C4 vertebra as a reference point. Then, the average movement distance was calculated and adopted.
Vertebral artery cerebral blood flow velocity | day 1 before any intervention, day 11, and day 60
  The ultrasound diagnostic device was used to measure the internal diameter of the vertebral artery. The sample volume was then positioned at the center of the vessel and the angle between the ultrasound beam and the blood flow direction was kept within 60°. The Color Doppler ultrasound examination was performed to measure the mean blood flow velocity of the vertebral artery by continuously observing 10 cycles.
Vertebral artery internal diameter | day 1 before any intervention, day 11, and day 60
  The ultrasound diagnostic device was used to measure the internal diameter of the vertebral artery. The sample volume was then positioned at the center of the vessel and the angle between the ultrasound beam and the blood flow direction was kept within 60°.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Study Chair — Site Coordinator of United Medical Group
Locations (6):
- China (6):
  - zhongshan affiliated No.1 Hospital, Guandong
  - HLJ older people hospital, Heilongjiang
  - Lankao Renmen Hospital, Henan
  - NY zhongxin Hospital, Naning
  - People's Hospital of SN tequ, Suzhu
  - Department of rehabilitation medicine, the first ZU hospital north campus, Zhenzhou